CLINICAL TRIAL: NCT02185716
Title: Comparison Of Ultrasound Guided Transversus Abdominis Plane Block (TAP) and Local Infiltration Analgesia During Laparoscopic Cholecystectomy Surgery
Brief Title: Transversus Abdominis Plane Block (TAP) for Laparoscopic Cholecystectomy Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, gulbin sezen, assistant of professor, Duzce University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-414
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Cholecystectomy, Laparoscopic; Pain, Postoperative
Keywords: Transversus abdominis plane block; levobupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Care Provider, Investigator

ARMS (3):
- local infiltration (Active Comparator): Group L (n=25) will be given total 30 ml 0.25 % levobupivacaine infiltration around trocar-site with injector in sterilized conditions without administering TAP block at the end of the operation
  Interventions: Drug: Levobupivacaine 0.5%
- Control (No Intervention): Only routine general anesthesia will be applied
- TAP (Experimental): Group T (n=25) will be given bilateral total 30 ml 0.25 % levobupivacaine administering TAP block under the guidance of ultrasound at the preoperative period.
  Interventions: Drug: Levobupivacaine 0.25 %

INTERVENTIONS:
Drug: Levobupivacaine 0.25 %
  Other Names: chirocaine
  Arms: TAP
Drug: Levobupivacaine 0.5%
  Other Names: chirocaine
  Arms: local infiltration

SUMMARY:
Postoperative pain is a significant cause of increased morbidity in the perioperative period, leading to patient discomfort and greater hospital length of stay. Laparoscopic cholecystectomy associated with significant postoperative pain, a substantial component of which is derived from abdominal wall incisions. Ultrasound-guided TAP block increasingly has been used for providing pain relief following abdominal surgery. We designed this study with the hypothesis that, administering TAP block with levobupivacaine in laparoscopic cholecystectomy provides superior analgesic effects than port-side infiltration.

DETAILED DESCRIPTION:
In this randomized and double-blind study, 75 patients, American Society of Anesthesiology (ASA) I-II risk group, between the ages of 20-60, who will undergo elective laporoscopic cholecystectomy operation under general anesthesia will be accepted. The patients will be divided into three groups and they will be given postoperative pain treatment with patient-controlled analgesia device. In hours of postoperative 1, 2, 4, 8, 12, 16 and 24, Visual analog scale (VAS) I (superficial pain), VAS II (deep pain), postoperative total analgesic proportion, nausea and vomiting, evaluation postoperative sedation score will be recorded (as conscious:0, asleep:1, deep sleep:2 ) in hours of postoperative 1, 2, 4, 8, 12, 16 and 24.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II risk group,
* between the ages of 20-60,
* undergo elective laporoscopic cholecystectomy operation under general anesthesia

Exclusion Criteria:

* allergy to anesthetic medication,
* coronary artery patients,
* obese patients,
* emergencies,
* pregnants,
* abdomen operation history
* heart block

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
postoperative pain scores | 24 hours
  VAS I (superficial pain), VAS II (deep pain) recorded in hours of postoperative 1, 2, 4, 8, 12, 16 and 24 h,

SECONDARY OUTCOMES:
postoperative total analgesic consumption | Postoperatively 24 h

OTHER OUTCOMES:
side effects | postoperatively 24 h
  In hours of postoperative 1, 2, 4, 8, 12, 16 and 24 nausea, and vomiting will be recorded.Nausea (0=non-existent, 1=mild, 2 = severe) and vomiting (0=non-existent, 1=mild, 2 = severe) of the patients will be scored postoperatively on a 3-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gülbin Sezen, MD,PhD, Principal Investigator — Duzce University
Locations (1):
- Duzce University Medical Faculty, Düzce, Turkey (Türkiye)

REFERENCES:
- [Result] Wassef M, Lee DY, Levine JL, Ross RE, Guend H, Vandepitte C, Hadzic A, Teixeira J. Feasibility and analgesic efficacy of the transversus abdominis plane block after single-port laparoscopy in patients having bariatric surgery. J Pain Res. 2013 Nov 27;6:837-41. doi: 10.2147/JPR.S50561. eCollection 2013. PMID 24348067
- [Result] Keir A, Rhodes L, Kayal A, Khan OA. Does a transversus abdominis plane (TAP) local anaesthetic block improve pain control in patients undergoing laparoscopic cholecystectomy? A best evidence topic. Int J Surg. 2013;11(9):792-4. doi: 10.1016/j.ijsu.2013.05.039. Epub 2013 Jun 11. PMID 23770342